CLINICAL TRIAL: NCT05671081
Title: Dexmedetomidine Versus Magnesium Sulfate in Ultrasound Guided Bilateral Bi-level Erector Spinae Plane Block in Corrective Scoliosis Surgery: A Randomized Controlled Clinical Trial.
Brief Title: Dexmedetomidine Versus Magnesium Sulfate in Ultrasound Guided Bilateral Bi-level Erector Spinae Plane Block in Corrective Scoliosis Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R263/2022
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia , Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Magnesium Sulfate; Narcotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anethesia +Dexmedetomidine plus Bupivacaine for Erector spinae plane block (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- General anethesia +Magnesium sulfate plus Bupivacaine for Erector spinae plane block (Active Comparator)
  Interventions: Drug: Magnesium sulfate
- general anesthesia+conventional postoperative narcotic analgesia (Active Comparator)
  Interventions: Drug: Narcotic Analgesics

INTERVENTIONS:
Drug: Dexmedetomidine — patients will receive combined general anesthesia and bilateral bilevel at T5 &T10 Erector spinae plane block with 20mL of bupivacaine 0.125 %. plus 0.5 μg/kgof Dexmedetomidine for each injection
  Arms: General anethesia +Dexmedetomidine plus Bupivacaine for Erector spinae plane block
Drug: Magnesium sulfate — patients will receive combined general anesthesia and bilateral bilevel at T5 &T10 Erector spinae plane block with 20mL of bupivacaine 0.125 %. plus 2 mg/kg Magnesium sulfate for each injection
  Arms: General anethesia +Magnesium sulfate plus Bupivacaine for Erector spinae plane block
Drug: Narcotic Analgesics — patients will receive general anesthesia and conventional intraoperative and postoperative analgesia
  Arms: general anesthesia+conventional postoperative narcotic analgesia

SUMMARY:
Posterior spinal fusion for scoliosis surgery may lead to severe postoperative pain which requires significant opioid use for adequate perioperative analgesia. This postoperative pain extends the time of recovery, and thus, safe, and efficient methods for perioperative analgesia are crucial and advantageous for early recovery and ambulation.

Traditional opioid-based analgesia techniques are characterized by well-known complications such as vomiting, nausea, sedation, and pruritus. Although regional anesthesia is an essential part of multimodal analgesia, available options are limited. Recently, an ultrasound (US)-guided erector spinae plane block (ESPB) method that anesthetizes ventral and dorsal rami of spinal nerves was introduced for the treatment of both postoperative and neuropathic pain.

Due to the arousing interest of several physicians, ESPB application is reported to be effective in the breast, weight loss, and lumbosacral spine surgeries as it reduces the need for analgesic drugs. The main advantages of the ESPB are technical simplicity, minimal risk for the spinal cord, and fewer complications.

The ESP block is a fascial plane block that aims to inject a local anesthetic mixture within a plane beneath the erector spinae muscle at the transverse process of the vertebra. ESP block can provide effective postoperative analgesia for upper abdominal surgery when performed at the thoracic vertebra 7-8 level. ESP block acts probably by diffusion of local anaesthetic into the paravertebral space. The advantages of ESP block are its ease of performance and safety. Owing to its superficial location, away from vessels and nerves, the complications associated with paravertebral block can be avoided.

The effect of magnesium was first recognized for the treatment of arrhythmia and preeclampsia, and its effect on anaesthesia and analgesia has recently been recognized. Magnesium sulphate has also been used as an adjunct to anaesthesia in recent years. It is also an effective analgesic agent for perioperative pain. Research has also reported that the intraoperative use of magnesium is characterized by a reduced use of anesthetics and muscle relaxants. Furthermore, opioid use, postoperative nausea and vomiting, hypertension, and shivering have met a decreased trend with the use of magnesium sulphate.

Magnesium sulfate (MgSO4) may be helpful as an analgesic adjuvant in regional anesthesia because it improves and prolongs the analgesic effect of local anesthetics; moreover, MgSO4 alone modulates the transmission of nociceptive stimuli and pain perception by blocking the N-methyl-D-aspartate (NMDA) receptor.

Dexmedetomidine (DE) is a potent α2 adrenoreceptor agonist and it is highly selective for α2 adrenoreceptor seven times more than clonidine. Many studies documented a prolonged duration and rapid onset of sensory block with the perineural injection of DE. Dexmedetomidine has been introduced as an adjuvant to local anaesthetics in both neuroaxial and peripheral nerve blocks. perineural dexmedetomidine has shown to prolong the duration of postoperative analgesia in addition to reducing the opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* patients who will be scheduled for indicated open corrective scoliosis surgery in the prone position.
* physical status American Society of Anesthesiologists (ASA) I or II.

Exclusion Criteria:

* patients refuse to participate.

  . -ASA physical status >II.
* patients who have contraindications to regional analgesic procedures as infection at injection site
* patients who have major illnesses (e.g., cardiac, respiratory, renal, hepatic or neurological).
* allergy to the study drugs
* a known history of recent opioid use
* obesity (body mass index (BMI) > 35 kg/m2)
* those who underwent revision surgery
* coagulopathy
* drug or alcohol abuse
* epilepsy, or a psychiatric illness that would interfere with the perception and assessment of pain.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
First time to analgesic requirement | 1st 48 hour
  All patients will receive an IV PCA system (Accufuser M8P, 100 mL: Woo Young Meditech Co, S. Korea). PCA was prepared with 100 mL of isotonic saline containing 50 mg morphine, and the selected system was adjusted to infuse a 5 mL bolus dose with a lockout interval of 15 minutes while the basal flow rate was switched off.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt